CLINICAL TRIAL: NCT00733174
Title: Rosiglitazone Therapy In The Prevention Of Coronary Artery Disease In Patients With Impaired Glucose Tolerance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Denver Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Jane Reusch, MD, Denver Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101797; COMIRB NO: 03-755
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Impaired Glucose Tolerance
Keywords: IGT
MeSH Terms: conditions — Glucose Intolerance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Rosiglitazone
  Interventions: Drug: Rosiglitazone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — tablet
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Subjects with impaired glucose tolerance will be randomized to either rosiglitazone or placebo for a 18 month period. The study will look at baseline, 12 month and 18 month data for exercise tolerance, coronary artery calcification and diabetes indicators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign the informed consent to participate in the study.
* Male or female adults ages 25-75 years.
* Female subjects must be postmenopausal (i.e., > 6 months without menstrual period), surgically sterile, or using effective barrier contraceptive measures (Intra-Uterine Device (IUD), diaphragm with spermicide or condom with spermicide).
* Women of childbearing potential must use effective barrier contraceptive measures for at least 1 month prior to visit 1, and should continue to use the same contraceptive method during the study and for 30 days after discontinuing study medication.
* Female subjects of childbearing potential must have a negative urine pregnancy test.
* Subjects must have an FPG < 126 mg/dL at Screening 1 AND Screening 2, a C-peptide > 2.0 ng/mL and a HbA1c <6.5%.
* Subjects must have a Body Mass Index 25-40 (must be < 300 lbs).
* Subjects must have a 2 hour post-prandial glucose 140-199 mg/dL at Screening 1 AND Screening 2. If the 2 hour post-prandial glucose result is 130-139 mg/dL at Screening 2, subjects will be allowed to repeat the OGTT.

Exclusion Criteria:

* Women who are lactating, pregnant, or planning to become pregnant during the study will be excluded.
* Women using hormone contraception or on hormone replacement therapy will be excluded.
* Subjects with any clinically significant abnormality identified on the Screening physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study will also be excluded.
* Use of any other investigational agents or participation in any other investigational studies during the study period will not be allowed.
* Patients will also be excluded if there is a presence of clinically significant hepatic disease or patient with LFT levels > 2 times the upper limit of normal laboratory range
* Subjects with a documented history of significant hypersensitivity (e.g., difficulty swallowing, difficulty breathing, tachycardia or skin reaction) to thiazolidinediones
* Subjects with any contraindications to rosiglitazone
* Presence of unstable or severe (New York Heart Association-NYHA class 3 or 4) angina, including angina requiring continual nitrate treatment for symptomatic relief, or coronary insufficiency
* Subjects with HYHA class 3 or 4 of congestive heart failure requiring drug therapy; systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg
* History of cancer (except non-melanomatous skin carcinoma)
* Active alcohol or drug abuse within the last 6 months
* Subjects with chronic diseases requiring periodic or intermittent treatment with oral or intravenous corticosteroids
* Subjects who are unable to understand dosing directions or swallow study medications
* Subjects who are currently smoking
* Subjects unable to adhere to protocol requirements.
* Persons with angina or any other cardiac or pulmonary symptoms that would potentially limit exercise performance will be excluded.
* Persons taking prescription or over-the-counter weight loss medications or persons on a weight loss program with ongoing weight loss, or starting an intensive exercise program within 30 days of screening will also be excluded.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-03; Primary Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Effect of rosiglitazone vs. placebo on exercise tolerance | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- South Federal Family Practice, Denver, Colorado, United States